CLINICAL TRIAL: NCT04318392
Title: Non-invasive Profiling of Breath Volatile Organic Compounds in Sarcoidosis: Relation to the Lung Microbiome and Markers of Disease Progression.
Brief Title: Breath Analysis in Patients With Suspected Sarcoidosis: The VOCs-IS Study
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B00081
Record Dates: First submitted 2019-04-08; First posted 2020-03-24 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Sarcoidosis
Keywords: Sarcoidosis; Volatile Organic Compounds; Breathomics
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis | interventions — Respiratory Physiological Phenomena; Blood Specimen Collection; Genetic Testing; Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma stored for metabolomic analysis. Blood stored for future genetic analysis (voluntary).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with suspected sarcoidosis: Patients presenting with suspected sarcoidosis.
  Interventions: Other: Breath Analysis; Other: Pulmonary Function Tests; Other: Blood sampling and storage for genetic analysis; Other: Blood sampling and storage of plasma for metabolomic analysis; Other: Bronchoalveolar lavage; Other: Sputum Culture
- Healthy controls: Healthy controls matched for age and gender. Recruitment of spouses and partners will also take place where possible.
  Interventions: Other: Breath Analysis; Other: Spirometry

INTERVENTIONS:
Other: Breath Analysis — Breath analysis using the ReCIVA device will take place during each study visit.
Other: Pulmonary Function Tests — Full Pulmonary Function Tests will be performed at baseline and during each study visit if not performed as part of routine clinical care.
  Groups: Patients with suspected sarcoidosis
Other: Blood sampling and storage for genetic analysis — Additional voluntary consent will be sought for blood sampling and storage for genetic analysis at baseline.
  Groups: Patients with suspected sarcoidosis
Other: Blood sampling and storage of plasma for metabolomic analysis — Blood sampling and storage of plasma for metabolomic analysis will take place during each study visit.
  Groups: Patients with suspected sarcoidosis
Other: Bronchoalveolar lavage — Bronchoalveolar lavage will be performed at baseline on all participants undergoing investigation with bronchoscopy or EBUS as part of routine clinical care for investigation of suspected sarcoidosis.
  Other Names: BAL
  Groups: Patients with suspected sarcoidosis
Other: Sputum Culture — Sputum will be collected during each study visit if the patient can spontaneously expectorate and will be sent for routine microbial analysis as well as metagenomic sequencing.
  Groups: Patients with suspected sarcoidosis
Other: Spirometry — Spirometry will be performed on all healthy controls prior to enrolment into the study
  Groups: Healthy controls

SUMMARY:
Sarcoidosis is a chronic condition which predominantly affects the lungs and lymph glands within the chest, however, may affect any organ within the body. At the present time, very little is known as to the exact cause of sarcoidosis and it is widely believed that the condition arises due to overreaction of the immune system to an unknown trigger in the environment such as an infection. Alongside this, the clinical course and progression of the condition varies considerably; some patients have a very mild form which does require any specific treatment, where as other patients develop a more severe form which can lead to permanent scarring (fibrosis) of the lungs if left untreated. At the present time it is difficult to predict how a patient will be affected by their sarcoidosis as there is a distinct lack of clinically useful markers which help predict prognosis and identify people at risk of disease progression or those who require treatment.

The main aims of this study are to use a technique which captures and analyses breath samples to provide a profile of the chemicals known as volatile organic compounds (VOCs) which are present in the exhaled breath of patients with sarcoidosis. Specifically the study would look to see if these VOCs are different in patients with sarcoidosis compared to people who do not have sarcoidosis or any lung conditions. In addition, the study would look to see how these breath profiles relate to potential infections, change over time or in response to treatment with steroids.

The study will involve a total of 80 patients presenting with suspected sarcoidosis and involve a total of four study visits over the course of twelve months. During each study visit a sample of breath will be collected alongside a blood test to look for markers of disease activity as well as completion of two questionnaires relating to a patients degree of breathlessness and quality of life. At the start of the study an additional questionnaire will be completed to identify possible risk factors for the development of sarcoidosis as well as the option of providing a sample of blood for genetic testing (which is voluntary). In patients undergoing a bronchoscopy or endobronchial ultrasound (EBUS), a sample of fluid which naturally lines the airways (bronchoalveolar lavage) will also be taken and used for metagenomic sequencing to try and identify any microbes which might be present within the lung and airways.

DETAILED DESCRIPTION:
Sarcoidosis is chronic condition which can affect any organ within the body, however frequently involves the lungs and thoracic lymph nodes. The exact cause of the disease remains uncertain and it is thought that the immune system overreacts to a possible inhaled antigen in the environment. A role has been suggested for triggers such as certain types of infection.

The clinical course and prognosis of sarcoidosis is extremely variable. Some patients make a full recovery without the need for any specific treatment, however up to a third of patients may develop a more severe form of the disease which can lead to scarring and fibrosis of the lungs. As such, the treatment of sarcoidosis focuses on suppressing the immune system, however the evidence to support this remains weak. Furthermore, such treatment may place the patient at risk of long-term side effects.

At the present time, there is a lack of useful markers which not only help diagnose the condition, but also help to predict and identify those patients at risk of developing more severe disease or who may require treatment.

The purpose of this study is to use a technique which analyses breath samples to provide a profile of chemicals which are present in the exhaled breath of patients with sarcoidosis. It is important to know if this profile differs from healthy people, relates to infections or changes over time, particularly in response to treatment. As such, hopefully this technique will provide an alternative way of monitoring the disease or predicting progression.

This is an observational case-control study of patients with suspected sarcoidosis receiving standard care at two NHS hospitals over the course of 12 months. At baseline, if patients are undergoing a bronchoscopy or endobronchial ultrasound and lymph node biopsy as part of their routine clinical care an additional sample of bronchoalveolar lavage fluid will be collected and used for metagenomic sequencing to identify the presence of any infections such as bacterial, viruses or fungi. In addition, patients will also be invited to provide additional voluntary consent for an extra biopsy to be taken which would also be used for metagenomic sequencing. Alongside this a sample of breath would be collected using the ReCIVA device (Owlstone Medical, Cambridge, UK), as well as blood sampling and storage for biomarker analysis. Patients would also be asked to complete three questionnaires including the medical research council dyspnoea score (MRC) and King's Sarcoidosis Health Related Quality of Life Questionnaire (KSQ) relating to their employment, level of breathlessness, symptoms and quality of life. Additional voluntary consent would also be sought for an extra blood test to be taken at baseline and stored for future genetic analysis.

During the course of study, three further follow-up visits would then take place at 3, 6 and 12 months. During each visit a sputum sample would be collected (if the patient was able to expectorate spontaneously) as well as repeated blood and breath sampling and completion of the medical research council dyspnoea score and King's Sarcoidosis Questionnaire. Pulmonary function tests would be performed as part of routine clinical care. At the end of the study, a repeat high resolution computerised tomography (CT) scan of the chest would take place to look for any new changes related to sarcoidosis and assess the activity of the disease.

The study will aim to recruit a total of 80 patients presenting with suspected sarcoidosis across both sites. In a subset of 10 participants, repeated breath sampling will take place two weeks from baseline to assess for reproducibility.

Alongside patients with suspected sarcoidosis, 40 healthy volunteers (including partners or spouses) will be recruited for breath sampling at baseline.

The study is being undertaken as part of a PhD programme and is funded by a grant from British Lung Foundation. Ethical approval has been granted from the North West - Greater Manchester Central Research Ethics Committee (IRAS Number 241100).

ELIGIBILITY:
Participants with Suspected Sarcoidosis:

Inclusion Criteria:

* Age >18 years
* Suspected pulmonary sarcoidosis undergoing investigations for diagnosis, staging and treatment consideration or discussion at a designated interstitial lung disease multidisciplinary meeting (this includes participants with stage I disease characterised by the presence of hilar or mediastinal lymphadenopathy)

Exclusion Criteria:

* Significant respiratory co-morbidity where the primary major respiratory diagnosis is not sarcoidosis
* Current smoker or ex-smoker (having ceased smoking <3 months duration)
* Extra-pulmonary sarcoidosis without any evidence of pulmonary involvement (characterised by normal pulmonary function tests and no radiological evidence of thoracic sarcoidosis on HRCT or chest radiography)
* Inability to provide written consent
* Self-reported lower respiratory tract infection, or treatment with antibiotics for a lower respiratory tract infection or any other infection within the previous 4 weeks

Healthy Volunteers:

Inclusion Criteria:

* Age >18 - 70 years
* Normal spirometry

Exclusion Criteria:

* Current smoker or ex-smoker (having ceased smoking <3 months duration)
* History of uncontrolled diabetes, respiratory, inflammatory gastroenterological, autoimmune or renal disease (characterised by an eGFR <30ml/min/1.73m2)
* Self-reported lower respiratory tract infection, or treatment with antibiotics for a lower respiratory tract infection or any other infection within the previous 4 weeks
* Inability to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting with suspected sarcoidosis
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Baseline volatile organic compounds (VOCs) in breath samples in patients with sarcoidosis compared to healthy controls and in relation to the lung microbiome. | The start of the study.
  The investigators would like to determine if the VOC profile obtained in breath samples from patients with sarcoidosis is different from people who do not have the condition and furthermore to determine if this is related to any microbes which might be present within the lung microbiome.

SECONDARY OUTCOMES:
Baseline VOCs in relation to markers of disease progression over twelve months. | Twelve months.
  The investigators would like to determine if the VOC breath profile is different in patients who have evidence of disease progression which is indicated by changes in the forced vital capacity, changes on high resolution computerised tomography scan, medical research council dyspnoea score and King's sarcoidosis quality of life questionnaire scores over a period of twelve months.
Exhaled VOC profiles related to markers of steroid response. | Twelve months.
  The investigators would like to determine if the VOC breath profile differs in patients who receive treatment and those that do not over a period of twelve months.
Exhaled VOC profiles and reproducibility in sarcoidosis | Two weeks after starting the study.
  The investigators would like to determine if the breath profiles obtained in patient with sarcoidosis are able to be reproduced in those who undergo repeated breath sampling at two weeks after starting the study.
Exhaled VOC profiles related to potential microbial markers of disease including any bacterial or fungal agents present in tissue obtained during EBUS/transbronchial lung biopsy. | The start of the study.
  The investigators would like to determine if the VOC breath profile related to microbes which might be present within lymph node and lung tissue obtained in patients with suspected sarcoidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Fowler, MD FRCP, Principal Investigator — The University of Manchester
Locations (2):
- United Kingdom (2):
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich, Norfolk
  - Wythenshawe Hospital, Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Undecided